CLINICAL TRIAL: NCT03669419
Title: QoR-9 AS predicTor of postopErative Complications
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: QoR- ASPECT
Record Dates: First submitted 2018-08-06; First posted 2018-09-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Complications
Keywords: Outcome; Postoperative Complications; Failure to rescue; QoR-9; patient-centred questionnaire
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: QoR 9 Questionnaire — The QoR-9 as established patient-centred outcome measure, which is validated in German language, is surveyed preoperatively, as well as on postoperative day 1 and 3 after non-cardiac surgery. Postoperative complications are evaluated using the Clavien-Dindo Score. A follow-up is intended after 6 months. Preoperative risk is estimated using the ASA (American Society of Anesthesiologists) and the POSPOM (Preoperative Score to predict postoperative mortality) score.

SUMMARY:
Aim of the study is to evaluate, whether the self administered quality of recovery (QoR-9) questionnaire can predict postoperative complications after non-cardiac surgery and whether preoperative risk estimates can be improved by implementation of the QoR-9 as postoperative screening tool.

DETAILED DESCRIPTION:
The QoR-9 as established patient-centred outcome measure, which is validated in German language, is surveyed preoperatively, as well as on postoperative day 1 and 3 after non-cardiac surgery. We showed in a pilot study that this score reveals a high sensitivity to detect patients with a disturbed health status through a detailed and time-consuming physical examination.We want to evaluate if short screening tools can be used to categorize patients with increased risk for developing postoperative complicationsTherefore, patients undergoing non-cardiac surgery are informed preoperatively about the study and written informed consent is obtained. Afterwards, the QoR-9, as well as validated preoperative risk scores are obtained. Relevant intra- and immediate postoperative factors are recorded. On postoperative day 1 and 3 patients perform the QoR-9. Postoperative complications during hospital stay are determined using the Clavien Dindo score by searching the patients 'record. After 6 months the patients are contacted via telephone and the QoR-9 is obtained. 6-months mortality is determined.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* undergoing non-cardiac surgery
* good knowledge of German language

Exclusion Criteria:

* blind
* out-patient
* pregnant
* psychiatric disturbance that preclude cooperation
* decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3854 patients undergoing surgery at Klinikum Rechts der Isar, Technical University who have good knowledge of German Language.
  Surgical procedures include all departments except cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3854 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-07-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Complications evaluated by Clavien- Dindo Score | Date of Surgery till Discharge from Hospital (approximately 30 days)
  Nine domains are evaluated: Pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, wound, haematological and pain. Each domain is graded between grade I and V (death of a patient).

SECONDARY OUTCOMES:
hospital mortality | Date of Surgery till Discharge from Hospital (approximately 30 days)
  Rate of Mortality among study patients
6-month mortality | 6 month after date of surgery
  Mortality among patients 6 months after surgery
Superiority of QoR-9 questionnaire against common Outcome Score | Date of surgery until 6 month follow-up
  Comparison of different risk estimates and Outcome Scores

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jungwirth, Prof., Study Director — Department of Anesthesia, Klinikum rechts der Isar, TU Munich
Locations (1):
- Klinikum Rechts der Isar, Technische Universität München, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Result] Anetsberger A, Blobner M, Krautheim V, Umgelter K, Schmid S, Jungwirth B. Self-Reported, Structured Measures of Recovery to Detect Postoperative Morbidity. PLoS One. 2015 Jul 24;10(7):e0133871. doi: 10.1371/journal.pone.0133871. eCollection 2015. PMID 26207620
- [Result] Myles PS, Grocott MP, Boney O, Moonesinghe SR; COMPAC-StEP Group. Standardizing end points in perioperative trials: towards a core and extended outcome set. Br J Anaesth. 2016 May;116(5):586-9. doi: 10.1093/bja/aew066. No abstract available. PMID 27106961
- [Result] Ghaferi AA, Birkmeyer JD, Dimick JB. Variation in hospital mortality associated with inpatient surgery. N Engl J Med. 2009 Oct 1;361(14):1368-75. doi: 10.1056/NEJMsa0903048. PMID 19797283
- [Result] Regenbogen SE, Ehrenfeld JM, Lipsitz SR, Greenberg CC, Hutter MM, Gawande AA. Utility of the surgical apgar score: validation in 4119 patients. Arch Surg. 2009 Jan;144(1):30-6; discussion 37. doi: 10.1001/archsurg.2008.504. PMID 19153322
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542